CLINICAL TRIAL: NCT02136914
Title: Efficacy and Safety of ADS-5102 (Amantadine HCl) Extended Release Capsules for the Treatment of Levodopa Induced Dyskinesia in Parkinson's Disease Patients (EASE LID Study)
Brief Title: ADS-5102 for the Treatment of Levodopa Induced Dyskinesia (EASE LID Study)
Acronym: EASE LID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADS-AMT-PD301
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Dyskinesia; Levodopa Induced Dyskinesia (LID); Parkinson's Disease
Keywords: Levodopa Induced Dyskinesia; LID; Parkinsonism
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADS-5102 (Experimental): ADS-5102 (amantadine HCl extended release)
  Interventions: Drug: ADS-5102
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADS-5102 — Oral capsules to be administered once nightly at bedtime, for 25 weeks
  Other Names: amantadine HCl extended release
  Arms: ADS-5102
Other: Placebo — Oral capsules to be administered once nightly at bedtime, for 25 weeks
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, 2-arm, parallel group study to evaluate the efficacy and safety of ADS-5102 extended release (ER) capsules, an investigational formulation of amantadine, dosed once nightly at bedtime for the treatment of levodopa induced dyskinesia (LID) in subjects with Parkinson's disease (PD). The novel pharmacokinetic profile of ADS-5102 is expected to achieve i) maximal concentrations in the early morning through mid-day, when LID can be troublesome, and ii) lower concentrations in the evening, potentially reducing the negative impact of amantadine on sleep. This pharmacokinetic profile could enable higher doses to be tolerated with a once-nightly ER formulation than can be tolerated with an immediate-release formulation. The once-nightly dosing regimen may also provide enhanced convenience and compliance.

In a previous clinical study, ADS-5102 met its primary endpoint; LID was significantly reduced as measured by the change in UDysRS score over 8 weeks vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB/REB/IEC-approved informed consent form
* Parkinson's disease, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria
* On a stable regimen of antiparkinson's medications for at least 30 days prior to screening, including a levodopa preparation administered not less than three times daily, and willing to continue the same doses and regimens during study participation
* Following diary training, the subject is willing and able to understand and complete the 24-hour PD home diary (caregiver/study partner assistance allowed)
* Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and subject must be willing to continue the same doses and regimens during study participation (this criterion does not apply to medications that are being taken pre-study only on an as-needed basis)

Exclusion Criteria:

* History of neurosurgical intervention related to Parkinson's disease (e.g. deep brain stimulation)
* History of seizures within 2 years prior to screening
* History of stroke or transient ischemic attack (TIA) within 2 years prior to screening
* History of cancer within 5 years prior to screening, with the following exceptions: adequately treated non-melanomatous skin cancers, localized bladder cancer, non-metastatic prostate cancer or in situ cervical cancer
* Presence of cognitive impairment, as evidenced by a Mini-Mental Status Examination (MMSE) score of less than 24 during screening
* If female, is pregnant or lactating
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize an effective method of contraception from screening through at least 4 weeks after the completion of study treatment.
* Treatment with an investigational drug or device within 30 days prior to screening
* Treatment with an investigational biologic within 6 months prior to screening
* Current participation in another clinical trial

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Director, Study Director — Adamas Pharmaceuticals, Inc.
Locations (43):
- United States (40):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sun City, Arizona
  - Fountain Valley, California
  - Pasadena, California
  - Reseda, California
  - Sacramento, California
  - Torrance, California
  - Ventura, California
  - Aurora, Colorado
  - Manchester, Connecticut
  - Boca Raton, Florida
  - Gainesville, Florida
  - Naples, Florida
  - Port Charlotte, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Bingham Farms, Michigan
  - West Bloomfield, Michigan
  - Golden Valley, Minnesota
  - St Louis, Missouri
  - Albany, New York
  - Commack, New York
  - New York, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - Kirkland, Washington
  - Milwaukee, Wisconsin
- Canada (3):
  - Edmonton, Alberta
  - Toronto, Ontario
  - Regina, Saskatchewan

REFERENCES:
- [Derived] Hauser RA, Mehta SH, Kremens D, Chernick D, Formella AE. Effects of Gocovri (Amantadine) Extended-Release Capsules on Motor Aspects of Experiences of Daily Living in People with Parkinson's Disease and Dyskinesia. Neurol Ther. 2021 Dec;10(2):739-751. doi: 10.1007/s40120-021-00256-1. Epub 2021 May 22. PMID 34024025
- [Derived] Mehta SH, Pahwa R, Tanner CM, Hauser RA, Johnson R. Effects of Gocovri (Amantadine) Extended Release Capsules on Non-Motor Symptoms in Patients with Parkinson's Disease and Dyskinesia. Neurol Ther. 2021 Jun;10(1):307-320. doi: 10.1007/s40120-021-00246-3. Epub 2021 Apr 17. PMID 33864229
- [Derived] Elmer LW, Juncos JL, Singer C, Truong DD, Criswell SR, Parashos S, Felt L, Johnson R, Patni R. Pooled Analyses of Phase III Studies of ADS-5102 (Amantadine) Extended-Release Capsules for Dyskinesia in Parkinson's Disease. CNS Drugs. 2018 Apr;32(4):387-398. doi: 10.1007/s40263-018-0498-4. PMID 29532440
- [Derived] Pahwa R, Tanner CM, Hauser RA, Isaacson SH, Nausieda PA, Truong DD, Agarwal P, Hull KL, Lyons KE, Johnson R, Stempien MJ. ADS-5102 (Amantadine) Extended-Release Capsules for Levodopa-Induced Dyskinesia in Parkinson Disease (EASE LID Study): A Randomized Clinical Trial. JAMA Neurol. 2017 Aug 1;74(8):941-949. doi: 10.1001/jamaneurol.2017.0943. PMID 28604926

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 126 Participants with Parkinson's disease (PD) and Levodopa-induced Dyskinesia (LID) were randomized at 41 study sites in the United States and Canada. The first subject was randomized on 20 May 2014 and the last subject completed on 18 November 2015.
Pre-assignment Details: All randomized subjects who received ≥ 1 dose of study drug (123) were included in the Safety Analysis Population (60 placebo, 63 ADS-5102); all randomized subjects who received ≥ 1 dose of study drug and provided ≥ 1 postbaseline efficacy assessment (121) were included in the Modified Intent-to-Treat (MITT) population (58 placebo, 63 ADS-5102).
Groups:
- Placebo: Placebo: oral capsules administered once nightly at bedtime for 25 weeks
- ADS-5102 (340 mg): 340 mg dose of ADS-5102 (amantadine hydrochloride [HCl] extended release): oral capsules administered once nightly at bedtime for 25 weeks
Period: Overall Study
Arm/Group | Placebo | ADS-5102 (340 mg)
Started | 63 | 63
Received Study Drug | 60 | 63
Completed | 42 | 42
Not Completed | 21 | 21
Not completed — Sponsor's Decision to Stop the Study | 7 | 7
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Subject Unwilling to Proceed | 7 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Did Not Receive Study Drug | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Groups:
- ADS-5102 (340 mg): 340 mg dose of ADS-5102 (amantadine HCl extended release): oral capsules administered once nightly at bedtime for 25 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | ADS-5102 (340 mg) | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 32 | 59
  >=65 years | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.59) | 63.9 (9.43) | 64.7 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 37 | 35 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 51 | 60 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 53 | 60 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Unified Dyskinesia Rating Scale (UDysRS) [Mean (Standard Deviation); unit: units on a scale] — The UDysRS is a dyskinesia rating scale that evaluates involuntary movements associated with PD; the UDysRS consists of the following sub-parts: IA, IB, IIA, IIB, III, and IV. The total score is the sum of all individual sub-parts, and scores for this measure can range from 0-104. The total objective score is the sum of Part III (which measures objective impairment) and Part IV (which measures objective disability), and scores for this measure can range from 0-44. For both the total score and total objective score, a higher score indicates more severe PD.
  units on a scale
    Total Score | 38.2 (11.20) | 40.9 (13.34) | 39.6 (12.37)
    Total Objective Score (Parts III, IV) | 15.3 (6.66) | 16.4 (7.72) | 15.9 (7.21)
PD Home Diary [Mean (Standard Deviation); unit: hours] — A PD home diary was used to score 5 different conditions in 30-minute intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
  hours
    Asleep | 8.02 (1.446) | 7.78 (1.732) | 7.90 (1.597)
    Off | 2.94 (2.105) | 3.16 (2.372) | 3.05 (2.239)
    ON without Troublesome Dyskinesia | 8.59 (2.815) | 8.34 (3.466) | 8.46 (3.155)
    ON with Troublesome Dyskinesia | 4.46 (1.933) | 4.72 (2.537) | 4.59 (2.257)
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) [Mean (Standard Deviation); unit: units on a scale] — The MDS-UPDRS Parts I, II, III, and IV examined non-motor experiences of daily living, motor experiences of daily living, motor examination, and motor complications, respectively. Each Part contains items/questions, each rated on a scale from 0 (normal) to 4 (severe). The range of total scores for each Part is as follows: Part I, 0-52; Part II, 0-52; Part III, 0-132; Part IV, 0-24. Combined Parts I, II, and III is the sum of scores from Parts I, II, and III and has a scale range of 0-236. Parts 4.1 and 4.2 each has a scale range of 0-4. Higher scores indicate more severe PD. Population: For Part I and combined Parts I, II, and III, in the placebo group, the data is based on 59 patients only.
  units on a scale
    Part I: number analyzed (Participants) | 59 | 63 | 122
    Part I | 11.5 (4.17) | 12.5 (6.18) | 12.0 (5.31)
    Part II | 15.8 (5.80) | 15.7 (6.77) | 15.8 (6.29)
    Part III | 24.6 (12.10) | 25.9 (14.49) | 25.3 (13.34)
    Combined Parts I, II, and III: number analyzed (Participants) | 59 | 63 | 122
    Combined Parts I, II, and III | 51.9 (16.95) | 54.2 (20.37) | 53.1 (18.75)
    Part IV | 11.3 (2.36) | 11.8 (2.95) | 11.6 (2.68)
    Part IV, Item 4.1 | 2.4 (0.82) | 2.6 (0.94) | 2.5 (0.89)
    Part IV, Item 4.2 | 2.5 (0.54) | 2.6 (0.56) | 2.5 (0.55)
Time Since PD Diagnosis [Mean (Standard Deviation); unit: years] | 8.85 (3.911) | 9.45 (4.372) | 9.16 (4.148)
Duration of Levodopa Treatment [Mean (Standard Deviation); unit: years] | 6.82 (3.346) | 7.82 (3.719) | 7.33 (3.563)
Duration of LID [Mean (Standard Deviation); unit: years] | 3.21 (2.491) | 4.05 (3.085) | 3.64 (2.831)
Hoehn and Yahr Stage [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale, from 1-5, describes the patient's PD progression. The higher the score the more severe the symptoms of PD.
  units on a scale | 2.3 (0.56) | 2.2 (0.54) | 2.3 (0.55)
Subjects taking Antiparkinson Medication [Count of Participants; unit: Participants] — Patients may have been taking more than 1 antiparkinson medication at Baseline
  Participants
    Levodopa (Sinemet or Stalevo) | 60 | 63 | 123
    Dopamine Agonist | 34 | 29 | 63
    MAO Inhibitors | 24 | 26 | 50
    COMT Inhibitor | 9 | 7 | 16
    Anticholinergics | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Unified Dyskinesia Rating Scale (UDysRS) Score at Week 12
Description: The UDysRS is a dyskinesia rating scale from 0-104; it evaluates involuntary movements associated with PD. A higher score indicates more severe PD. The UDysRS was measured at Baseline and Weeks 2, 8, 12, 18, and 24.
Time Frame: Baseline to Week 12
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (340 mg)
Number analyzed (Participants) | 58 | 63
units on a scale | -8.0 (1.64) | -15.9 (1.62)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); 46 subjects per treatment arm provided 90% power using a 2-sided test at 5% significance; Test type: Superiority; p = 0.0009, Linear Mixed Model w/ Repeated Measures; Change from baseline is a dependent variable, treatment group is a factor, and the baseline value is a covariate; Least Squares Mean Difference = -7.9, 95% CI 2-sided [-12.5 to -3.3], Standard Error of Mean 2.30

2. Secondary Outcome: Change From Baseline in the Unified Dyskinesia Rating Scale (UDysRS) Score at Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (340 mg)
Number analyzed (Participants) | 58 | 63
units on a scale | -6.3 (1.94) | -15.6 (1.87)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0008, Linear Mixed Model w/ Repeated Measures; Least Squares Mean Difference = -9.3, 95% CI 2-sided [-14.7 to -4.0], Standard Error of Mean 2.70

3. Secondary Outcome: Change in the Standardized PD Home Diary (ON Time Without Troublesome Dyskinesia, ON Time With Troublesome Dyskinesia, OFF Time)
Description: A PD home diary was used to score 5 different conditions in 30-minute intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia. The results were based on 2 consecutive 24-hour diaries taken prior to the day of randomization and prior to the Week 2, 8, 12, 18, and 24 visits.
Time Frame: Baseline (BL) to Week 12 (W12) and Week 24 (W24)
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | ADS-5102 (340 mg)
Number analyzed (Participants) | 58 | 63
hours
  Change in ON time w/o troublesome dyskinesia (W12) | 0.82 (0.432) | 3.56 (0.434)
  Change in ON time w/o troublesome dyskinesia (W24) | 1.37 (0.456) | 3.59 (0.440)
  Change in OFF time (W12) | 0.32 (0.263) | -0.59 (0.265)
  Change in OFF time (W24) | 0.22 (0.282) | -0.58 (0.268)
  Change in ON time w/ troublesome dyskinesia (W12) | -1.58 (0.358) | -3.12 (0.359)
  Change in ON time w/ troublesome dyskinesia (W24) | -1.86 (0.380) | -3.31 (0.363)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p < 0.0001, Linear Mixed Model w/ Repeated Measures — Change from Baseline in ON time without troublesome dyskinesia at Week 12; Least Squares Mean Difference = 2.74, 95% CI 2-sided [1.53 to 3.96], Standard Error of Mean 0.612
Statistical Analysis 2: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0007, Linear Mixed Model w/ Repeated Measures — Change from Baseline in ON time without troublesome dyskinesia at Week 24; Least Squares Mean Difference = 2.22, 95% CI 2-sided [0.96 to 3.47], Standard Error of Mean 0.634
Statistical Analysis 3: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0171, Linear Mixed Model w/ Repeated Measures — Change from Baseline in OFF time at Week 12; Least Squares Mean Difference = -0.90, 95% CI 2-sided [-1.64 to -0.16], Standard Error of Mean 0.373
Statistical Analysis 4: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0406, Linear Mixed Model w/ Repeated Measures — Change from Baseline in OFF time at Week 24; Least Squares Mean Difference = -0.81, 95% CI 2-sided [-1.58 to -0.04], Standard Error of Mean 0.389
Statistical Analysis 5: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0031, Linear Mixed Model w/ Repeated Measures — Change from Baseline in ON time with troublesome dyskinesia at Week 12; Least Squares Mean Difference = -1.54, 95% CI 2-sided [-2.55 to -0.53], Standard Error of Mean 0.508
Statistical Analysis 6: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.0072, Linear Mixed Model w/ Repeated Measures — Change from Baseline in ON time with troublesome dyskinesia at Week 24; Least Squares Mean Difference = -1.45, 95% CI 2-sided [-2.49 to -0.40], Standard Error of Mean 0.526

4. Secondary Outcome: Change in the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Combined Score (Parts I, II, and III)
Description: The MDS-UPDRS Parts I, II, and III examined non-motor experiences of daily living, motor experiences of daily living, and motor examination, respectively. Each Part contains items or questions that were each rated on a scale from 0 (normal) to 4 (severe). The Combined Parts I, II, and III (representing the sum of the individual scores from Parts I, II, and III) has a scale range of 0-236. Higher scores, whether for individual Parts or the sum of the combined Parts, indicate more severe PD.
Time Frame: Baseline (BL) to Week 12 (W12) and Week 24 (W24)
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (340 mg)
Number analyzed (Participants) | 58 | 63
units on a scale
  Change from BL at Week 12 | -4.0 (1.96) | -5.2 (1.92)
  Change from BL at Week 24 | -3.5 (2.60) | -1.3 (2.45)
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.6833, Linear Mixed Model w/ Repeated Measures — Change from Baseline in MDS-UPDRS at Week 12; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-6.6 to 4.3], Standard Error of Mean 2.74
Statistical Analysis 2: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.5557, Linear Mixed Model w/ Repeated Measures — Change from Baseline in MDS-UPDRS at Week 24; Least Squares Mean Difference = 2.1, 95% CI 2-sided [-5.0 to 9.2], Standard Error of Mean 3.58

5. Secondary Outcome: Clinician's Global Impression of Change (CGI-C) in Overall PD Symptoms
Description: The CGI-C consisted of a single question that assessed the investigator's global impression of the subject's change from Baseline in overall PD symptoms, including but not limited to LID. The CGI-C required that the investigator rate the extent to which the subject's PD had improved or worsened (from marked worsening to marked improvement). The CGI-C was assessed at Baseline and Weeks 2, 8, 12, 18, and 24.
Time Frame: Baseline to Week 12 and Week 24
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ADS-5102 (340 mg)
Number analyzed (Participants) | 58 | 63
Participants
  Week 12: Marked Improvement | 2 | 18
  Week 12: Moderate Improvement | 9 | 20
  Week 12: Minimal Improvement | 10 | 13
  Week 12: No Change | 25 | 9
  Week 12: Minimal Worsening | 10 | 2
  Week 12: Moderate Worsening | 2 | 0
  Week 12: Marked Worsening | 0 | 1
  Week 24: number analyzed (Participants) | 54 | 62
  Week 24: Marked Improvement | 5 | 14
  Week 24: Moderate Improvement | 10 | 17
  Week 24: Minimal Improvement | 12 | 12
  Week 24: No Change | 17 | 7
  Week 24: Minimal Worsening | 6 | 5
  Week 24: Moderate Worsening | 4 | 5
  Week 24: Marked Worsening | 0 | 2
Statistical Analysis 1: Comparison: ADS-5102 (340 mg); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Baseline to Week 12
Statistical Analysis 2: Comparison: ADS-5102 (340 mg); Test type: Superiority; p = 0.1071, Cochran-Mantel-Haenszel — Baseline to Week 24

ADVERSE EVENTS:
Time Frame: Baseline through Week 25
Arm/Group | Placebo | ADS-5102 (340 mg)
All-Cause Mortality (participants affected / at risk) | 0/60 | 1/63
Serious Adverse Events (participants affected / at risk) | 3/60 | 7/63
Other Adverse Events (participants affected / at risk) | 36/60 | 56/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | ADS-5102 (340 mg) (N=63)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ON and OFF phenomenon (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | ADS-5102 (340 mg) (N=63)
Hallucination, any type (Psychiatric disorders) | 1 | 18
Hallucination, visual (Psychiatric disorders) | 1 | 15
Hallucination, auditory (Psychiatric disorders) | 0 | 5
Oedema peripheral (General disorders) | 0 | 15
Dizziness (Nervous system disorders) | 0 | 14
Dry mouth (Gastrointestinal disorders) | 0 | 11
Constipation (Gastrointestinal disorders) | 3 | 9
Fall (Injury, poisoning and procedural complications) | 5 | 10
Urinary tract infection (Infections and infestations) | 5 | 7
Anxiety (Psychiatric disorders) | 1 | 6
Contusion (Injury, poisoning and procedural complications) | 1 | 6
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 6
Abnormal dreams (Psychiatric disorders) | 2 | 4
Depression (Psychiatric disorders) | 1 | 4
Headache (Nervous system disorders) | 2 | 4
Balance disorder (Nervous system disorders) | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No